CLINICAL TRIAL: NCT05676099
Title: TSC Alliance Tuberous Sclerosis Complex (TSC) Biosample Repository and Natural History Database
Brief Title: TSC Biosample Repository and Natural History Database
Status: Recruiting | Type: Observational
Sponsor: National Tuberous Sclerosis Association (Other)
Responsible Party: Sponsor
Other Study IDs: 15039
Record Dates: First submitted 2022-12-21; First posted 2023-01-09 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Tuberous Sclerosis; Lymphangioleiomyomatosis
MeSH Terms: conditions — Tuberous Sclerosis; Lymphangioleiomyomatosis | interventions — Phlebotomy; Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Biological materials will be collected at different timepoints in conjunction with procedures that are done for clinical reasons or when consent is given to collect the sample expressly for this research study. Historical cord blood, dried blood spot or placental tissue samples may be collected. Postmortem organ tissue may be collected with consent from the parent/legal guardian of the deceased person with TSC who was enrolled in this protocol or from whom medical records are available to enter relevant clinical data in the NHD.
  Blood spots may be collected using at-home commercial devices shipped to participants or at CSS using available resources. Blood spots may be created when blood samples arrive at VAI. Biosamples may be processed and analyzed for genetic variants using whole genome sequencing (WGS) or other sequencing methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Phlebotomy — Participants may elect to submit a blood sample to the Biosample Repository.
Procedure: Buccal (cheek) swab — Participants may elect to submit a buccal swab sample to the Biosample Repository.
Genetic: Genetic Testing — Biosamples may be processed and analyzed for genetic variants using whole genome sequencing (WGS) or other sequencing methods. Participants whose samples are processed in this manner may be contacted and provided the option to receive TSC1 or TSC2 genetic variant results by opting in using Consent to Return of Genetic Results Form. Participants will be offered a one-time genetic counseling session to review their results, free of charge. CLIA-certified, TSC1 or TSC2 genetic variant results will be returned to participants who opt in to receive such results. Additionally, negative results and results not able to be clinically certified will also be offered to participants with a one-time genetic counseling session to review their results, free of charge using the Return of Genetic Research Results Template Letter. CSS will be responsible for informing clinic participants that their samples have been sequenced and offer to connect participant to the TSC Alliance for further information.
Other: Tissue donation after routine clinical procedure — Participants may elect to submit a tissue sample to the Biosample Repository following a medical procedure.

SUMMARY:
The TSC Biosample Repository collects and stores samples of blood, DNA, and tissues that scientists can request to use in their research. The samples we collect are all linked to clinical data in the TSC Natural History Database. The TSC Natural History Database captures clinical data to document the impact of the disease on a person's health over his or her lifetime. This data may be collected retrospectively or prospectively.

DETAILED DESCRIPTION:
The purpose of the project which is sponsored by the TSC Alliance is to learn more about tuberous sclerosis complex (TSC) which may lead to new treatments for conditions that affect different areas of the body such as the brain, kidney, heart, lungs, and skin. The TSC Alliance TSC Biosample Repository (BSR) was established to provide a central biobank at the Van Andel Institute (VAI) Biorepository in Grand Rapids, Michigan for the collection of blood, tissues, and cells from a vast number of individuals with TSC.

The TSC Alliance Natural History Database (NHD), established in 2006, will serve as the central repository of de-identified clinical data associated with biosamples collected from individuals with TSC. The NHD research project involves collection of retrospective and prospective private information on individuals with a diagnosis of TSC over their lifespan (i.e., a longitudinal study). The VAI Biorepository will distribute biosamples and NHD data to researchers as approved by the TSC Alliance.

This project also aims to collect biosamples and clinical data on people affected by sporadic lymphangioleiomyomatosis (sporadic LAM). LAM is a common symptom reported in TSC that may occur outside the context of a TSC diagnosis (i.e., sporadic LAM patients).

The collection of biosamples will be at a clinical study site (CSS) such as a TSC Alliance recognized TSC clinic, a non-CSS such as a participant's home, an educational meeting, or by other clinical partners (CP) with institutional review board (IRB) approval of this protocol and informed consent forms. Collection of biosamples may also occur at a non-CSS or by a licensed phlebotomist (e.g., via partnership with mobile phlebotomy companies). The VAI Biorepository will provide collection kits, instructions, and materials to the CSS, non-CSS, CP, or directly to participant.

The CSS, CP, non-CSS, or authorized representative will ship collected biosamples to the VAI Biorepository for processing and storage according to their IRB-approved standard operating procedures. The VAI Biorepository will distribute biosamples to investigators as approved by the TSC Alliance. Their accreditation under the Biorepository Accreditation Program of the College of American Pathologists (CAP) will stand as the governing rules for best practices. Distribution of biosamples will require receipt of the investigator's IRB approval and a material transfer agreement (MTA) executed between the approved investigator and the TSC Alliance.

Clinical data in the NHD associated with a biosample will be provided to an investigator as approved by the Natural History Database-Biosample Repository (NHD-BSR) Steering Committee.

This project is open to individuals of all ages with a diagnosis of tuberous sclerosis complex or lymphangioleiomyomatosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of tuberous sclerosis complex or lymphangioleiomyomatosis (sporadic LAM).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An individual must have a diagnosis of tuberous sclerosis complex, based on the current clinical and genetic diagnostic criteria. The individual may enroll if they have a diagnosis of sporadic LAM. All persons with tuberous sclerosis complex are eligible to participate, such as individuals with limited decisional capacity.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Natural History data and biosamples including blood, tissue, or other types of biological samples from individuals with TSC | Average 15 years
  The purposes of this project are to:
  * Collect biosamples such as blood, tissue, fluid, or other types of bodily samples from people with TSC.
  * Collect information about people with TSC over their lifetime.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Roberds, PhD, Principal Investigator — TSC Alliance
Locations (24):
- United States (22):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Loma Linda University Children's Hospital, Loma Linda, California
  - University of California Los Angeles, Los Angeles, California
  - Jack & Julia Center for TSC, Oakland Children's Hospital and Research Center, Oakland, California
  - The Children's Hospital, Denver, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Chicago Comer Children's Hospital Neurogenetic Clinic, University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - TSC Alliance, Silver Spring, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minnesota Epilepsy Group, Roseville, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Scottish Rite Hospital for Children, Dallas, Texas
  - Texas Childrens Hospital Baylor College of Medicine, Houston, Texas
  - Memorial Hermann-Texas Medical Center (University of Texas Houston), Houston, Texas
  - Children's National Medical Center, Fairfax, Virginia
- Canada (2):
  - Centre Hospitalier de L'Université de Montréal (Chum), Montreal
  - Sainte-Justine Université de Montréal, Montreal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pounders AJ, Rushing GV, Mahida S, Nonyane BAS, Thomas EA, Tameez RS, Gipson TT. Racial differences in the dermatological manifestations of tuberous sclerosis complex and the potential effects on diagnosis and care. Ther Adv Rare Dis. 2022 Dec 10;3:26330040221140125. doi: 10.1177/26330040221140125. eCollection 2022 Jan-Dec. PMID 37180419
- [Background] Rubtsova VI, Chun Y, Kim J, Ramirez CB, Jung S, Choi W, Kelly ME, Lopez ML, Cassidy E, Rushing G, Aguiar DJ, Lau WL, Ahdoot RS, Smith M, Edinger AL, Lee SG, Jang C, Lee G. Circulating biomarkers of kidney angiomyolipoma and cysts in tuberous sclerosis complex patients. iScience. 2024 Jun 13;27(7):110265. doi: 10.1016/j.isci.2024.110265. eCollection 2024 Jul 19. PMID 39027368
- [Background] Parthasarathy S, Mahalingam R, Melchiorre J, Harowitz J, Devinsky O. Mortality in tuberous sclerosis complex. Epilepsy Behav. 2021 Aug;121(Pt A):108032. doi: 10.1016/j.yebeh.2021.108032. Epub 2021 Jun 1. PMID 34087679
- [Background] Chivukula S, Modiri O, Kashanian A, Babayan D, Ibrahim GM, Weil AG, Tu A, Wu JY, Mathern GW, Fallah A. Effect of Gene Mutation on Seizures in Surgery for Tuberous Sclerosis Complex. Can J Neurol Sci. 2021 May;48(3):327-334. doi: 10.1017/cjn.2020.185. Epub 2020 Aug 28. PMID 32854808
- [Background] Gupta A, de Bruyn G, Tousseyn S, Krishnan B, Lagae L, Agarwal N; TSC Natural History Database Consortium. Epilepsy and Neurodevelopmental Comorbidities in Tuberous Sclerosis Complex: A Natural History Study. Pediatr Neurol. 2020 May;106:10-16. doi: 10.1016/j.pediatrneurol.2019.12.016. Epub 2020 Feb 4. PMID 32139167
- [Background] Song J, Swallow E, Said Q, Peeples M, Meiselbach M, Signorovitch J, Kohrman M, Korf B, Krueger D, Wong M, Sparagana S. Epilepsy treatment patterns among patients with tuberous sclerosis complex. J Neurol Sci. 2018 Aug 15;391:104-108. doi: 10.1016/j.jns.2018.06.011. Epub 2018 Jun 15. PMID 30103955
- [Background] Jeong A, Nakagawa JA, Wong M. Predictors of Drug-Resistant Epilepsy in Tuberous Sclerosis Complex. J Child Neurol. 2017 Dec;32(14):1092-1098. doi: 10.1177/0883073817737446. PMID 29129154
- [Background] Jeong A, Wong M. Systemic disease manifestations associated with epilepsy in tuberous sclerosis complex. Epilepsia. 2016 Sep;57(9):1443-9. doi: 10.1111/epi.13467. Epub 2016 Jul 15. PMID 27417921
- [Background] Kothare SV, Singh K, Hochman T, Chalifoux JR, Staley BA, Weiner HL, Menzer K, Devinsky O. Genotype/phenotype in tuberous sclerosis complex: associations with clinical and radiologic manifestations. Epilepsia. 2014 Jul;55(7):1020-4. doi: 10.1111/epi.12627. Epub 2014 Apr 22. PMID 24754401
- [Background] Kothare SV, Singh K, Chalifoux JR, Staley BA, Weiner HL, Menzer K, Devinsky O. Severity of manifestations in tuberous sclerosis complex in relation to genotype. Epilepsia. 2014 Jul;55(7):1025-9. doi: 10.1111/epi.12680. Epub 2014 Jun 10. PMID 24917535
- [Background] van Eeghen AM, Nellist M, van Eeghen EE, Thiele EA. Central TSC2 missense mutations are associated with a reduced risk of infantile spasms. Epilepsy Res. 2013 Jan;103(1):83-7. doi: 10.1016/j.eplepsyres.2012.07.007. Epub 2012 Aug 3. PMID 22867869
- [Background] Ehninger D, Sano Y, de Vries PJ, Dies K, Franz D, Geschwind DH, Kaur M, Lee YS, Li W, Lowe JK, Nakagawa JA, Sahin M, Smith K, Whittemore V, Silva AJ. Gestational immune activation and Tsc2 haploinsufficiency cooperate to disrupt fetal survival and may perturb social behavior in adult mice. Mol Psychiatry. 2012 Jan;17(1):62-70. doi: 10.1038/mp.2010.115. Epub 2010 Nov 16. PMID 21079609
- [Background] Boggarapu S, Roberds SL, Nakagawa J, Beresford E. Characterization and management of facial angiofibroma related to tuberous sclerosis complex in the United States: retrospective analysis of the natural history database. Orphanet J Rare Dis. 2022 Sep 14;17(1):355. doi: 10.1186/s13023-022-02496-2. PMID 36104799
- [Background] Aronow ME, Nakagawa JA, Gupta A, Traboulsi EI, Singh AD. Tuberous sclerosis complex: genotype/phenotype correlation of retinal findings. Ophthalmology. 2012 Sep;119(9):1917-23. doi: 10.1016/j.ophtha.2012.03.020. Epub 2012 May 16. PMID 22608477
- [Background] Mowrey K, Northrup H, Rougeau P, Hashmi SS, Krueger DA, Ebrahimi-Fakhari D, Towbin AJ, Trout AT, Capal JK, Franz DN, Rodriguez-Buritica D. Frequency, Progression, and Current Management: Report of 16 New Cases of Nonfunctional Pancreatic Neuroendocrine Tumors in Tuberous Sclerosis Complex and Comparison With Previous Reports. Front Neurol. 2021 Apr 9;12:627672. doi: 10.3389/fneur.2021.627672. eCollection 2021. PMID 33897589
- [Background] Swallow E, King S, Song J, Peeples M, Signorovitch JE, Liu Z, Prestifilippo J, Frost M, Kohrman M, Korf B, Krueger D, Sparagana S. Patterns of Disease Monitoring and Treatment Among Patients With Tuberous Sclerosis Complex-related Angiomyolipomas. Urology. 2017 Jun;104:110-114. doi: 10.1016/j.urology.2017.02.036. Epub 2017 Mar 2. PMID 28263820
- [Background] Hsieh LS, Wen JH, Nguyen LH, Zhang L, Getz SA, Torres-Reveron J, Wang Y, Spencer DD, Bordey A. Ectopic HCN4 expression drives mTOR-dependent epilepsy in mice. Sci Transl Med. 2020 Nov 18;12(570):eabc1492. doi: 10.1126/scitranslmed.abc1492. PMID 33208499
- [Background] Giannikou K, Martin KR, Abdel-Azim AG, Pamir KJ, Hougard TR, Bagwe S, Tang Y, MacKeigan JP, Kwiatkowski DJ, Henske EP, Lam HC. Spectrum of germline and somatic mitochondrial DNA variants in Tuberous Sclerosis Complex. Front Genet. 2023 Jan 30;13:917993. doi: 10.3389/fgene.2022.917993. eCollection 2022. PMID 36793390
- [Background] Bhaoighill MN, Falcon-Perez JM, Royo F, Tee AR, Webber JP, Dunlop EA. Tuberous Sclerosis Complex cell-derived EVs have an altered protein cargo capable of regulating their microenvironment and have potential as disease biomarkers. J Extracell Vesicles. 2023 Jun;12(6):e12336. doi: 10.1002/jev2.12336. PMID 37337371
- [Background] Loubert F, House AA, Larochelle C, Major P, Keezer MR. Development and internal validation of a clinical risk score to predict incident renal and pulmonary tumours in people with tuberous sclerosis complex. J Med Genet. 2024 Sep 24;61(10):943-949. doi: 10.1136/jmg-2023-109717. PMID 38977299
- See also: TSC Alliance Webpage for Biosample Repository and Natural History Database — https://www.tscalliance.org/get-involved/participate-in-research/tsc-biosample-repository-and-natural-history-database/